CLINICAL TRIAL: NCT05847621
Title: Linking Individuals Needing Care for Substance Use Disorders in Urban Emergency Departments to Peer Coaches (LINCS UP): RCT Component
Brief Title: Linking Individuals Needing Care for Substance Use Disorders to Peer Coaches
Acronym: LINCS UP: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joseph Carpenter, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005553; R01CE003509 (NIH); 2025P009769 (Other: Emory IRB)
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person peer recovery coaching with linkage to recovery resources (Experimental): PRCs will meet patients at bedside (in person). They will also schedule and perform follow up calls after the participant is discharged from the ED to provide ongoing support and facilitate re-linkage to recovery resources, if needed.
  Follow-up data collection on day 7, 30, 90 post discharge.
  Interventions: Behavioral: Peer recovery coaching with linkage to recovery resources
- Telemedicine-based peer recovery coaching with linkage to recovery resources (Experimental): PRCs will meet patients via a tablet-based video call (telemedicine). They will also schedule and perform follow up calls after the participant is discharged from the ED to provide ongoing support and facilitate re-linkage to recovery resources, if needed.
  Follow-up data collection on day 7, 30, 90 post discharge.
  Interventions: Behavioral: Peer recovery coaching with linkage to recovery resources
- Usual Care (Active Comparator): Participants in the usual care arm will be provided with a list of community recovery resources. No callbacks or re-linkage to recovery resources.
  Follow-up data collection on day 7, 30, 90 post discharge.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Peer recovery coaching with linkage to recovery resources — Peer recovery coach (PRC) assessment of the participant's state of change, engage in motivational interviewing techniques, and link the participant to community-based recovery resources according to the needs of the participant. They will also schedule and perform follow up calls after the participant is discharged from the ED to provide ongoing support and facilitate re-linkage to recovery resources, if needed.
  Arms: In-person peer recovery coaching with linkage to recovery resources; Telemedicine-based peer recovery coaching with linkage to recovery resources
Behavioral: Usual Care — Participants will be provided with a list of community recovery resources.
  Arms: Usual Care

SUMMARY:
This is a 3-arm randomized controlled trial. Participants will be randomized via a maximally tolerated imbalance randomization procedure using NCI's Clinical Trial Randomization Tool with 1:1:1 allocation to each group: in-person peer recovery coaching (PRC) with linkage to recovery resources, telemedicine-based peer recovery coaching with linkage to recovery resources, or usual care.

In the PRC arms, PRCs will meet patients at bedside (in person) or via a tablet-based video call (telemedicine). They will assess the participant's state of change, engage in motivational interviewing techniques, and link the participant to community-based recovery resources according to the needs of the participant. They will also schedule and perform follow up calls after the participant is discharged from the ED to provide ongoing support and facilitate re-linkage to recovery resources, if needed.

Participants in the usual care arm will be provided with a list of community recovery resources, but there will be no PRC interaction or direct linkage to resources through the study.

Follow up visits will take place at 7, 30, and 90 days after enrollment. Most will take place via telephone, but participants will be given the option of an in-person visit if they so desire.

DETAILED DESCRIPTION:
Deaths from drug overdose have risen to record levels since the onset of the COVID-19 pandemic, disproportionately impacting Black individuals and people experiencing homelessness. Fewer than one-third of the 8.3 million individuals living with an illicit drug use disorder in 2019 reported receiving treatment. Telemedicine services have increased access to care for many patients living with substance use disorders (SUD), but the long-term role of this treatment approach in SUD care is uncertain. Multifaceted strategies are needed to build recovery capital and link vulnerable individuals to recovery resources.

Emergency department (ED) visits are an opportunity to screen for SUDs, initiate treatment, and link to recovery resources. Observational studies have noted that consultation with a peer recovery coach (PRC) was well-received in EDs, with high rates of engagement and satisfaction. PRCs facilitate conversations allowing patients to express their ideal pathway to recovery, provide linkage to services across the social ecology, and follow up to support recovery, including re-linkage to resources as needed. Nonetheless, their role in ED screening and linkage to resources, including the potential role of telemedicine, has not been rigorously evaluated.

The investigators will conduct a randomized controlled trial enrolling 600 subjects across three arms: in-person peer coaching with linkage to recovery support services and callbacks, telemedicine-based peer coaching with linkage and callbacks, or usual care. Results will inform other EDs considering a peer recovery coach program for patients presenting with SUD-related conditions. By utilizing telemedicine, this model will be rapidly scalable and readily implemented at other facilities.

ELIGIBILITY:
Inclusion Criteria:

1. ED patient or hospitalized through the ED within last 24 hours
2. Age 18 years or older
3. Able to speak and understand English
4. Clinically sober, able to provide informed consent
5. Score of 3 or greater - "moderate level", "substantial level", or "severe level" of problems related to drug abuse - on Drug Abuse Screening Test (DAST-10).(103, 104)
6. Willing to follow study procedures and complete research follow-up calls
7. Have at least one reliable contact number

Exclusion Criteria:

1. Medically or psychiatrically unstable as determined by treating physician
2. Prisoner or in police custody
3. Prior participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in number of participants with successful linkage to at least one recovery resource | Baseline, 30 and 90 days after enrollment
  Change in number of participants with successful linkage to at least one recovery resource (formal addiction treatment, Recovery Community Organization (RCO), or harm reduction organization) at 30 days and 90 days after enrollment.

SECONDARY OUTCOMES:
Change in Brief Assessment of Recovery Capital (BARC-10) | Baseline, 7, 30, and 90 days after enrollment
  This outcome will be evaluated obtaining a score on a scale. The range of possible responses is 10-60. Higher score correlates with better outcome.
Change in number of successful engagements with PRC after ED visit | Baseline, 7, 30, and 90 days after enrollment
  Change in number of successful engagements with PRC (peer recovery coach) after ED visit
Change in number of episodes of re-linkage to recovery resources | Baseline, 7, 30, and 90 days post intervention
  Change in number of episodes of re-linkage to recovery resources
Self-reported substance use in last 30 days | Baseline, 30 and 90 days post intervention
  Self-reported substance use in last 30 days as measured by Timeline Follow-back (TLFB). It will be reported in number of episodes per day.
Number of fatal overdose events | 90 days post intervention
  Number of fatal overdose events will be collected
Number of nonfatal overdose events | 90 days post intervention
  Number of nonfatal overdose events will be collected
Number of Emergency Department (ED) visits | 90 days post intervention
  Number of ED visits will be collected
Number of hospitalizations | 90 days post intervention
  Number of hospitalizations will be collected
Change in employment status | 90 days post intervention
  Choices include: disabled, employed 32 hours or more per week, employed less than 32 hours per week, full-time student, homemaker, on medical leave, only temporarily laid off/sick leave/maternity leave, other, part-time student, retired, unemployed, and unknown. This outcome would measure a change in employment status from any of the choices to another one.
Change in number of participants based on Housing status | Baseline, 7, 30, and 90 days post intervention
  Housing status will be reported specifying one of the categories: apartment, Single family house, homeless, shelter, dormitory, multifamily house. Number of participants will be reported in each category at 0, 7, 30, 90 days post intervention.
Change in Social connections and isolation score | Baseline, 7, 30, 90 days post intervention
  Social isolation scores range from 0 to 4, with 0 representing the highest level of social isolation and 4 representing the lowest level.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Carpenter, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be initiated upon written request to the PI and would ultimately be shared via a secure portal such as Microsoft OneDrive.
  Deidentified data files, the data dictionary, and the final protocol will be uploaded to the Emory Dataverse, which is a long-term repository offered through a partnership between Emory and the Odum Institute at the University of North Carolina and Chapel Hill. This repository has policies and procedures in place that will provide data access to qualified researchers, fully consistent with federal data sharing policies and applicable laws and regulations. Datasets are uniquely named with a persistent digital object identifier (DOI), and are downloadable directly through a web-based interface. Additional data documentation and de-identified data will be deposited for sharing along with data consistent with applicable laws and regulations. Submitted data will confirm with relevant data and terminology standards.
Supporting Information: Study Protocol
Time Frame: Data sharing will be initiated upon written request to the PI and would ultimately be shared via a secure portal such as Microsoft OneDrive.
  The investigators will make data publicly available within 30 months of completing data collection.
Access Criteria: Written request to the PI.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT05847621/ICF_000.pdf